CLINICAL TRIAL: NCT03661112
Title: A Pilot Study to Explore the Feasibility and Operational Pathways of Incorporating a Wrist-based Blood Pressure Monitoring Device Into the All of Us Research Program
Brief Title: Wrist-based Blood Pressure Monitoring Study
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Evan Muse, MD, PhD, Director, Digital Medicine, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: IRB-18-7119
Record Dates: First submitted 2018-05-03; First posted 2018-09-07 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Blood Pressure
Keywords: blood pressure; mobile device

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All of Us Research Program (AoURP) consortium members

SUMMARY:
To observe blood pressure variation in various real-world settings

DETAILED DESCRIPTION:
This is an observational study, which will utilize a wrist-based blood pressure monitor to explore blood pressure variation in up to 75 participants in various real-world settings. There is no intervention in this study. The study will take place over a 4-week period. During this time, participants will be asked to sample their blood pressures 1) at random times, several times per day; 2) during specific periods of either emotional stress or relaxation; 3) during guided orthostatic testing. Study participants will utilize an application on their smartphones to log the device-measured blood pressures and flag selected blood pressure measurements as either being part of the orthostatic testing or during periods of emotional stress/relaxation. At the close of the study a post-study questionnaire will be sent electronically to each participant.

ELIGIBILITY:
Inclusion Criteria:

* Consortium members within the All of Us Research Program
* ≥18 years of age
* Own an iOS or Android device

Exclusion Criteria:

* Inability to give informed consent
* <18 years of age
* Inability to understand written English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the All of Us Research Program (AoURP) Participant Center consortium (age > 18 years)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurements | 4 weeks
  The primary endpoint for this study is assessing variability in blood pressure measurements (both systolic and diastolic). Blood pressure measurements will be sought over the course of 4 weeks during the following activities:
  1. During waking hours (several times a day for at least 2 days out of the week)
  2. Orthostatic maneuvers (seated and then 1 minute after standing up)
  3. At times of stress and relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Evan D Muse, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Ben-Dov IZ, Kark JD, Ben-Ishay D, Mekler J, Ben-Arie L, Bursztyn M. Predictors of all-cause mortality in clinical ambulatory monitoring: unique aspects of blood pressure during sleep. Hypertension. 2007 Jun;49(6):1235-41. doi: 10.1161/HYPERTENSIONAHA.107.087262. Epub 2007 Mar 26. PMID 17389258
- [Background] Staessen JA, Thijs L, Fagard R, O'Brien ET, Clement D, de Leeuw PW, Mancia G, Nachev C, Palatini P, Parati G, Tuomilehto J, Webster J. Predicting cardiovascular risk using conventional vs ambulatory blood pressure in older patients with systolic hypertension. Systolic Hypertension in Europe Trial Investigators. JAMA. 1999 Aug 11;282(6):539-46. doi: 10.1001/jama.282.6.539. PMID 10450715
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Shimbo D, Abdalla M, Falzon L, Townsend RR, Muntner P. Role of Ambulatory and Home Blood Pressure Monitoring in Clinical Practice: A Narrative Review. Ann Intern Med. 2015 Nov 3;163(9):691-700. doi: 10.7326/M15-1270. Epub 2015 Oct 13. PMID 26457954
- [Background] Dolan E, Stanton A, Thijs L, Hinedi K, Atkins N, McClory S, Den Hond E, McCormack P, Staessen JA, O'Brien E. Superiority of ambulatory over clinic blood pressure measurement in predicting mortality: the Dublin outcome study. Hypertension. 2005 Jul;46(1):156-61. doi: 10.1161/01.HYP.0000170138.56903.7a. Epub 2005 Jun 6. PMID 15939805
- [Background] Steinhubl SR, Muse ED, Barrett PM, Topol EJ. Off the cuff: rebooting blood pressure treatment. Lancet. 2016 Aug 20;388(10046):749. doi: 10.1016/S0140-6736(16)31348-4. No abstract available. PMID 27560266